CLINICAL TRIAL: NCT04243031
Title: A Non-interventional, Prospective Clinical Performance Study of the QuantiFERON Access Kit to Demonstrate Clinical Accuracy Compared to a CE-marked In-Vitro Diagnostic Medical Device, in Participants With Varying Risk Factors for TB Infection and Disease.
Brief Title: QuantiFERON Access Clinical Performance Study Protocol
Status: Withdrawn | Type: Observational
Why Stopped: Business Decision
Sponsor: QIAGEN Gaithersburg, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: TMF-17-1056-1
Record Dates: First submitted 2020-01-23; First posted 2020-01-27 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Tuberculosis (TB)
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All subjects: Those with TB and those without TB.
  Interventions: Device: QFT Access

INTERVENTIONS:
Device: QFT Access — Measure of Interferon Gamma

SUMMARY:
Approximately 225 samples, obtained from participants with varying risk factors for TB infection and disease, will be tested using the QFT Access Kit and the comparator device QFT-Plus.

ELIGIBILITY:
Inclusion Criteria:

* 1. Be ≥ 18 years of age,
* 2. Have received no TB treatment or received treatment for less than 14 consecutive days.
* 3. Provide Informed Consent.

Exclusion Criteria:

* 1. They do not meet the inclusion criteria,
* 2. Blood handling was not completed using QFT-Plus
* 3. Incubation was <16 and >24 hours
* 4. Improperly collected and/or stored samples per Instructions For Use

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants coming to clinic
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2020-08-01 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
TB Result | At time of enrollment
  QFT Access result compared to the QFT-Plus result (positive, negative)

IPD SHARING:
Plan to Share IPD: No